CLINICAL TRIAL: NCT02590380
Title: A Randomized Controlled Trial: Comparison of a Top Loading MESA® Spinal System With MESA Rail™ and a Side Locking Pedicle Screw System for the Treatment of Adolescent Paediatric Spine Deformity
Brief Title: Comparing Pedicle Screw Systems for the Treatment of Adolescent Paediatric Spine Deformity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not started
Sponsor: K2M, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAS-029
Record Dates: First submitted 2015-10-22; First posted 2015-10-29 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent; paediatric; pediatric; scoliosis; spine deformity
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (MESA) (Active Comparator): Patients randomized to the treatment group will receive surgery with the MESA Rail Deformity System.
  Interventions: Device: MESA Rail Deformity System
- control group (USS II) (Active Comparator): Patients randomized to the control group will receive surgery with the DePuy Synthes USS II System.
  Interventions: Device: DePuy Synthes USS II System

INTERVENTIONS:
Device: MESA Rail Deformity System — The spinal deformity will be correction via a standard of care procedure performed by the principal investigator. The correction will be fixated with the MESA Rail Deformity System.
  Other Names: MESA Rail, K2M MESA Rail, MESA, K2M MESA
  Arms: treatment group (MESA)
Device: DePuy Synthes USS II System — The spinal deformity will be correction via a standard of care procedure performed by the principal investigator. The correction will be fixated with the DePuy Synthes USS II system.
  Other Names: DePuy, DePuy Synthes, Synthes, USS II, Universal Stainless
  Arms: control group (USS II)

SUMMARY:
Evaluation of the efficacy of the K2M MESA Rail™ Deformity System at improving coronal and sagittal correction of the adolescent idiopathic spine deformity in comparison to the side loading DePuy Synthes USS II pedicle screw system.

DETAILED DESCRIPTION:
Evaluation of the efficacy of the K2M MESA Rail™ Deformity System at improving coronal and sagittal correction of the adolescent idiopathic spine deformity in comparison to the side loading DePuy Synthes USS II pedicle screw system. This is a single-center, single-surgeon randomized controlled trial with follow-up evaluations of patients conducted at initial follow-up (2 weeks to 8 weeks), 3 months, 12 months and 24 months post-procedure. Adverse events will be monitored continuously.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Adolescent Idiopathic Scoliosis (AIS) with no associated syndrome requiring surgical treatment for selective thoracic/lumbar fusion with a minimum of five (5) instrumented vertebrae between T1-S1 as confirmed by patient history and radiographic studies. AIS cases must be classified as a Lenke type 1 or type 2 curve. No cervical vertebrae are to be incorporated into the construct.
2. Willingness and ability to comply with the requirements of the protocol including follow-up requirements.
3. Willing and able to sign a study specific informed consent form or, in the case of a patient who is a minor, provide assent and the minor patient's parent/legal guardian provides written consent to participate.
4. Age range of ≥ 11 years old and ≤ 21 years old at time of surgery.

Exclusion Criteria:

1. Previous anterior or posterior spine surgery at the index levels.
2. Previous posterior spine surgery (e.g., posterior element decompression) that destabilizes the cervical/thoracic/lumbar spine.
3. Active systemic infection or infection at the operative site.
4. Any sign of any spinal dysrhaphism (any cord abnormality).
5. Co-morbid medical conditions of the spine or upper/lower extremities that may affect the thoracic or lumbar spine neurological and/or pain assessment.
6. Metabolic bone disease such as osteoporosis that contradicts spinal surgery.
7. History of an osteoporotic fracture.
8. History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism.
9. Taking medications that may interfere with bony/soft tissue healing including chronic oral steroid use.
10. Known allergy to titanium or cobalt chrome.
11. Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia.
12. Insulin-dependent type 1 or type 2 diabetes.
13. Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion.
14. Pregnant, or intend to become pregnant, during the course of the study.
15. Severe obesity (Body Mass Index > 40).
16. Physical or mental condition (e.g., psychiatric disorder, senile dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain or quality of life.
17. Incarcerated at the time of study enrollment.
18. Current participation in an investigational study that may impact study outcomes.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Correction and Maintenance of Spinal Deformity (coronal) | Change from pre-operative to 3 months, 12 months and 24 months post-procedure
  Radiographic analysis of the spinal deformity in the coronal plane at the indicated time periods will be compared to the pre-operative measurements (OVERALL CHANGE from baseline at each timepoint). Later post-operative measurements will be compared to the initial correction values to establish maintenance of surgical correction over time.
Correction and Maintenance of Spinal Deformity (sagittal) | Change from pre-operative to 3 months, 12 months and 24 months post-procedure
  Radiographic analysis of the spinal deformity in the sagittal plane at the indicated time periods will be compared to the pre-operative measurements (OVERALL CHANGE from baseline at each timepoint). Later post-operative measurements will be compared to the initial correction values to establish maintenance of surgical correction over time.

SECONDARY OUTCOMES:
Back and Leg Pain 10cm Visual Analog Scale (VAS) | Initial follow-up (2 weeks to 8 weeks), 3 months, 12 months and 24 months post-procedure.
  The severity of back and leg pain will be evaluated in all study subjects using a 10-cm visual analog scale (VAS). The study will employ a 15% improvement for success. OVERALL CHANGE from baseline will be assessed at each timepoint.
SRS-22 | Initial follow-up (2 weeks to 8 weeks), 3 months, 12 months and 24 months post-procedure.
  Scoliosis and its treatment have a great impact on the quality of life of the affected patients. The Revised Scoliosis Research Society-22 (SRS-22r) is a specific questionnaire for spine conditions. It is applied to patients with idiopathic scoliosis, whose conditions and treatments have a great impact on their quality of life. The SRS-22r was created and revised with the purpose of evaluating this impact from the patient's point of view. The reviewed version contains 22 questions distributed into five domains: function/activity (FA), pain (P), self-image/appearance (SA), mental health (MH) and satisfaction with treatment (ST). The scores vary from 1 to 5, in which 5 is the best health quality of life of patients. OVERALL CHANGE from baseline will be assessed at each timepoint.
Estimated Blood Volume Loss/Salvage Return | Operative Data - to be collected immediately after case is completed. Estimated blood loss will be noted by the surgical/anesthesia team and this value can then be immediately collected.
  The amount of blood loss over the entire length of the surgery as well as salvage return volumes will be captured intraoperatively.
Length of Hospital Stay | At discharge (up to one week post surgery) - Once the subject has been released from the hospital, the length of hospital stay can be calculated using the intake and discharge dates.
  The length of hospital stay from the date of admission to the date of discharge will be calculated.
Return to Work/School | Initial follow-up (2 weeks to 8 weeks), 3 months, 12 months and 24 months post-procedure.
  The ability to and the time it takes for the subject to be cleared to return to work/school from the date of surgery will be documented. Once the subject has returned to the "baseline" status this question will not be asked.
Return to Sport/Physical Activity | Initial follow-up (2 weeks to 8 weeks), 3 months, 12 months and 24 months post-procedure.
  The ability to return to sport as performed by the individual patient pre operatively. Time to walking unaided, running, swimming, trampoline, contact sport, normal social interactions with peer group. Once the subject has returned to the "baseline" status this question will not be asked.
Use of Analgesia Post-Surgery | Initial follow-up (2 weeks to 8 weeks), 3 months, 12 months and 24 months post-procedure.
  The types and dosages of any analgesia taken by the patient post-surgery will be documented. Overall change from baseline (pre-operative medications) will be analyzed at each interval - anticipation is that use of analgesia decreases and/or ends after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, United Kingdom